CLINICAL TRIAL: NCT03053258
Title: Pilot Study to Evaluate Diagnostic Breath Analysis for Early Detection of Ventilator Acquired Pneumonia (VAP)
Brief Title: Diagnostic Breath Analysis for Detection of Ventilator Acquired Pneumonia (VAP)
Acronym: VAP-VOC
Status: Completed | Type: Observational
Sponsor: Landon Pediatric Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: Study 177 ZNose
Record Dates: First submitted 2017-02-09; First posted 2017-02-15 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Exhaled breath saved for re-test in thirty days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diagnostic Breath Analysis: VAP: Collection of exhaled breath samples
  Interventions: Device: Collection of exhaled breath sample

INTERVENTIONS:
Device: Collection of exhaled breath sample — Collect exhaled breath sample from patients with suspected VAP

SUMMARY:
Breath samples from patients with Ventilator Acquired Pneumonia (VAP) will be analyzed to identify Volatile Organic Compounds (VOC) that have been specifically associated with VAP in previous animal models.

Primary outcome measures will include the assessment of the zNose Diagnostic Breath Analysis System in the early detection of VOC's associated with VAP.

DETAILED DESCRIPTION:
On clinical suspicion of VAP, breath samples will be collected from the expiratory limb of the patient's ventilator tubing circuit. A sterile Tedlar collection bag will be used to connect to the sample port and collect the breath sample. The expiratory limb sample port will be utilized to ensure maintenance of the integrity of the ventilator circuitry. The breath samples will be analyzed via the ZNose breath analysis system.

Immediately following collection of breath samples, bronchoalveolar lavage fluid (BALF) will be collected and subjected to bacteriology testing for confirmation of VAP-positive and VAP-negative patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 48 hours of ventilation with suspected VAP infection. Suspicion of VAP infection based on clinical evaluation criteria:

  1. Three or more positive out of the following:

     1. Tympanic temperature > 38 °C or < 35.5 °C
     2. Blood leukocytosis (10,000/µl)
     3. More than ten leukocytes in Gram stain of tracheal aspirate (in high-flow field)
     4. Positive culture of tracheal aspirate
  2. New, persistent, or progressive infiltrate on chest radiograph

Exclusion Criteria:

Patients with pre-existing structural lung disease (COPD, asthma, lung cancer, etc.), thrombocytopenia (< 40,000/µL) and other coagulation abnormalities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated patients with suspected VAP infection
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Diagnostic Breath Analysis | 6 months
  Diagnostic analysis of Volatile Organic Compounds in exhaled breath samples These are compared to known compounds associated with sepsis in exhaled breath in septic rats, such as the oliphenones.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Landon, MD, Principal Investigator — Ventura County Medical Center
Locations (1):
- Ventura County Medical Center, Ventura, California, United States

IPD SHARING:
Plan to Share IPD: No